CLINICAL TRIAL: NCT03190824
Title: Open-label, Multi-center Phase IIa Study to Evaluate the Efficacy, Safety, and Immunological Response of OBP-301, Telomerase Specific Replication-competent Oncolytic Adenovirus in Patients With Unresectable Metastatic Melanoma
Brief Title: Evaluate Efficacy, Immunological Response of Intratumoral/Intralesional Oncolytic Virus (OBP-301) in Metastatic Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneos Health (Other)
Collaborators: Oncolys BioPharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL03001; Interventional (Other: Oncolys BioPharma Inc)
Record Dates: First submitted 2017-03-07; First posted 2017-06-19 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Melanoma Stage III; Melanoma Stage Iv
Keywords: melanoma; immunotherapy; immune oncology; loco regional therapy; adenovirus; oncolytic virus; unresectable; telomerase
MeSH Terms: conditions — Melanoma; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OBP-301 (Experimental): Eligible patients with unresectable Stage III and IV melanoma will receive up to 13 treatments of OBP 301 at a concentration of 1 × 1012 virus particles (VP)/mL for 24 weeks.
  Interventions: Drug: OBP-301

INTERVENTIONS:
Drug: OBP-301 — A novel, replication-competent Ad5 based adenoviral construct that incorporates a human telomerase reverse transcriptase gene (hTERT) promoter.
  Other Names: Telomelysin

SUMMARY:
Open-label, single-arm, multi-center, Phase IIa study to evaluate the efficacy, safety, and immunological response of OBP 301 in patients with unresectable/unresected metastatic melanoma. This proof of concept study will be undertaken in male and female patients with unresectable Stage III and IV melanoma. Patients with unresectable/unresected mucosal melanoma may be enrolled after consultation with the Medical Monitor.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of this study is to evaluate the overall tumor sites response (objective response rate [ORR]) to OBP-301 in both injected and noninjected lesions up to and including Week 24 in patients with unresectable/unresected Stage III and IV melanoma. The ORR is defined as the rate of complete response (CR) and partial response (PR) based on the modified immune-related response criteria (irRC) 1.0. The modification is to allow the identification of up to 10 cutaneous, subcutaneous, and/or lymph node tumor lesions and identify the lesions as target and nontarget lesions.

Secondary Objectives:

* To evaluate the ORR up to and including Week 24 in injected target lesions based on the modified irRC 1.0 and Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* To evaluate the ORR up to and including Week 24 in noninjected target lesions based on modified irRC 1.0 and RECIST 1.1
* To evaluate the ORR in both injected and noninjected target lesions at Week 12 based on the modified irRC 1.0 and RECIST 1.1
* To evaluate duration of response and time to response
* To evaluate progression free survival (PFS) at Week 24 and Week 48
* To evaluate overall survival (OS) at Week 24 and Week 48
* To evaluate the safety of OBP 301

Exploratory Objective (optional):

The optional exploratory objective of this study is to investigate the tumor immunological response in blood and tumor tissue following treatment with OBP-301.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed malignant melanoma at Screening that is unresectable/unresected Stage IIIB, IIIC, IIID or IV. Patients with unresectable mucosal melanoma may be enrolled after consultation with the Medical Monitor.
2. Patients must have received and failed or refused available therapy for unresectable/unresected Stage III or IV melanoma.
3. Patients must be ≥ 18 years of age.
4. At least 2 cutaneous, subcutaneous and/or lymph node target lesions that are greater or equal to 1 cm in the longest diameter. One of the cutaneous, subcutaneous and/or lymph node target lesions should be designated at Screening as a noninjected target lesion. Willing to have biopsy specimens taken at Screening and at Week 6.
5. Life expectancy of ≥ 6 months from the first OBP-301 treatment.
6. Karnofsky Performance Status Scale (KPS) score of ≥ 70.
7. Adequate organ function, hematologic status, coagulation status, kidney function, and liver function as follows:

   * Absolute neutrophils > 1,500/µL
   * Hemoglobin > 9 g/dL, without transfusion or hematopoietic growth factor
   * Platelets > 100,000/µL. Patients with ≤ 100,000 platelet count may be allowed into the study on a case-by-case basis after consultation with the Medical Monitor.
   * Serum creatinine < 2 × upper limit of normal (ULN)
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2 × ULN except for patients with known liver metastases, in which case aspartate transaminase or alanine transaminase may be ≤ 5.0 × ULN
   * Total bilirubin < 2.0 mg/dL (≤ 3.0 mg/dL for patients with known Gilbert's syndrome)
   * Serum lactate dehydrogenase (LDH) levels < 1.5 × ULN
8. Understand the study requirements and the treatment procedures, and is willing to comply with all specified follow-up evaluations, and provides written informed consent before any study-specific tests or procedures are performed.
9. Patients of reproductive potential must use effective contraception for the duration of the study and for 3 months (90 days) after the last administered injection of OBP-301. Effective contraception includes oral contraceptives, implantable hormonal contraception, double-barrier method or intrauterine device.

Exclusion Criteria:

1. Patients who have had administration of chemotherapy, target therapy, and/or immunotherapy within the last 4 weeks before the first OBP-301 administration.
2. Patients who have received other investigational medication within the last 4 weeks or a period of its 5 half-lives (whichever is shorter) before the first OBP-301 administration.
3. Patients who have had radiotherapy within the last 4 weeks before the first OBP-301 administration.
4. Effects of any other prior therapies not reverted to ≤ Grade 1 (or ≤ Grade 2 for alopecia and peripheral neuropathy).
5. Patients who have any liver metastases or visceral metastasis of ≥ 3 cm, plus evidence of progression meeting irRC 1.0 within 1 month before the first OBP-301 administration.
6. Patients with clinically active brain metastases. However, patients with previously currently stable brain metastases on medication (i.e., steroids and/or anti-seizure medications) may be enrolled after consultation with the Medical Monitor.
7. Patients known to have acute or chronic active hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV).
8. Patients diagnosed with additional malignancy within 3 years before the first OBP-301 administration with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cervical and/or breast cancers.
9. Patients requiring chronic systemic immunosuppressive medication including pharmacologic dose of glucocorticoids or cyclosporine should be evaluated by the Medical Monitor for enrollment eligibility.
10. Uncontrolled intercurrent illness including, but not limited to, uncontrolled diabetes, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/psychological incompetence, whereby in the opinion of the Investigator the patient is assessed as being unable to provide information, consent, or comply with the study requirements and procedures.
11. Patients who are pregnant or breastfeeding, or expecting to conceive or father children within the projected timeframe of the study, starting from the time of the Screening Visit through 3 months (90 days) after the last OBP-301 administration. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at each visit before administration of OPB-301. A female not of childbearing potential is one who has undergone bilateral oophorectomy or who has had no menses for 12 consecutive months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2021-06-24 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate objective response rate [ORR]) to OBP-301 in both injected and noninjected lesions | up to Week 24
  Objective response rate [ORR]) to OBP-301 in both injected and noninjected lesions in patients with unresectable/unresected Stage III and IV melanoma. The modification is to allow the identification of up to 10 cutaneous, subcutaneous, and/or lymph node tumor lesions and identify the lesions as target and nontarget lesions.

SECONDARY OUTCOMES:
Overall Response Rate at weeks 6, 12, 18, and 24 in the combined and individual injected lesions | Week 24 and Week 48
  ORR at Weeks 6, 12, 18, and 24 in the combined and the individual injected and noninjected target lesions according to the modified irRC v1.0 and RECIST 1.1.
Best Overall Response Rate at weeks 6, 12, 18, and 24 in injected and noninjected lesions | Week 24 and Week 48
  Best overall response rate (ORR in injected and noninjected target lesions) based on the modified irRC 1.0 and the RECIST 1.1.
Time to Treatment Response from start date to end date | Week 24 and Week 48
  Time to Treatment Response (TTR): the start date is the date of first treatment (Injection 1, Day 1) and the end date is the date of first documented response (CR or PR).
Duration of response of injected and noninjected lesions | Week 24 and Week 48
  Duration of response (injected and noninjected lesions): applies only to patients whose best overall response is CR or PR. The start date is the date of first documented response (CR or PR) and the end date is the date of first documented disease progression or the date of death due to underlying cancer.
Progression Free Survival at weeks 24 and 48 | Week 24 and Week 48
  PFS at Week 24 and Week 48
Overall Survival at weeks 24 and 48 | Week 24 and Week 48
  OS at Week 24 and Week 48
Safety of OBP-301 as assessed by incidence of AEs and SAEs | Through study completion
  Incidence of AEs and serious adverse events (SAEs) as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE; version 4.03). Changes in clinical laboratory parameters (serum chemistry, coagulation parameters, hematology, urinalysis) from Baseline.Vital signs. Physical examination. Electrocardiogram (ECG).
Safety of OBP-301 as assessed by changes in clinical laboratory parameters | Through study completion
  Changes in clinical laboratory parameters (serum chemistry, coagulation parameters, hematology, urinalysis) from Baseline.

OTHER OUTCOMES:
Exploratory Analysis (optional) | Through study completion
  Local and systemic immunological response

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Institution
Locations (1):
- Research Site, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No